CLINICAL TRIAL: NCT04135066
Title: Westlake Nutrition and Brain Health Study
Acronym: WEBRAIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Westlake University (Other)
Collaborators: Sun Yat-sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 20190901ZJS0010
Record Dates: First submitted 2019-10-13; First posted 2019-10-22 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-05

CONDITIONS: Aging
Keywords: Brain structure and function; Nutrition; Microbiome; Continuous blood glucose monitoring
MeSH Terms: interventions — Glucose Tolerance Test

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group A (RG-WG-OGTT) (Other): Starting on Day 1 with a continuous glucose monitoring (CGM) sensor, refined grain breakfasts (RG) are provided on Days 3 and 4, whole grain breakfasts (WG) are provided on Days 6 and 7, and an oral glucose tolerance test (OGTT) is conducted on Day 9. On other days during CGM activation, breakfast is unrestricted.
  Interventions: Other: Refine grain breakfast; Other: Whole grain breakfast; Other: Oral Glucose Tolerance test (75g 2-hour)
- Group B (WG-OGTT-RG) (Other): Starting on Day 1 with a continuous glucose monitoring (CGM) sensor, whole grain breakfasts (WG) are provided on Days 3 and 4, an oral glucose tolerance test (OGTT) is conducted on Day 6, and refined grain breakfasts (RG) are provided on Days 8 and 9. On other days during CGM activation, breakfast is unrestricted.
  Interventions: Other: Refine grain breakfast; Other: Whole grain breakfast; Other: Oral Glucose Tolerance test (75g 2-hour)
- Group C (OGTT-RG-WG) (Other): Starting on Day 1 with a continuous glucose monitoring (CGM) sensor, an oral glucose tolerance test (OGTT) is conducted on Day 3, refined grain breakfasts (RG) are provided on Days 5 and 6, and whole grain breakfasts (WG) are provided on Days 8 and 9. On other days during CGM activation, breakfast is unrestricted.
  Interventions: Other: Refine grain breakfast; Other: Whole grain breakfast; Other: Oral Glucose Tolerance test (75g 2-hour)

INTERVENTIONS:
Other: Refine grain breakfast — After wearing continuous glucose monitoring device (CGM) on baseline, participants will be provided with breakfast A on two consecutive days in a whoe 14-day monitoring period. The appearance of breakfast A is pseudorandom. Breakfast A contains white bread (100g) and milk powder (25g). Since lunch and dinner would serve as wash-out meals, participants will be free to choose food but provide a record of their diets.
  Other Names: Breakfast A
Other: Whole grain breakfast — After wearing CGM on baseline, participants will be provided with breakfast B on two consecutive days in a whoe 14-day monitoring period. The appearance of breakfast B is pseudorandom. Breakfast B contains plain oats (70g) and milk powder (25g). Since lunch and dinner would serve as wash-out meals, participants will be free to choose food but provide a record of their diets.
  Other Names: Breakfast B
Other: Oral Glucose Tolerance test (75g 2-hour) — 75 g pure glucose with 300 mL water per time per person is applied. In the following 3 hours, participants are advised to rest in a seated position, avoiding unnecessary walking or exercise. Energy-giving food items were still prohibited within this interval.

SUMMARY:
The Westlake Nutrition and Brain Study (WEBRAIN), a sub-study of the Guangzhou Nutrition and Health Study, is a prospective cohort study of residents in Guangzhou city. WEBRAIN aims to explore the links between diet, gut microbiome, and brain health in elderly individuals through comprehensive phenotyping, including continuous blood glucose monitoring for standardized test meals, objective physical activity measurement, and brain magnetic resonance imaging.

DETAILED DESCRIPTION:
The gut-brain axis is implicated in neurodegenerative diseases through various mechanisms, with diet and nutrition linked to both gut and brain health. However, most evidence comes from animal models or small-scale human studies.

The Westlake Nutrition and Brain Study (WEBRAIN) aims to investigate the relationships among diet, gut microbiome, and brain structure and function in a large human cohort through comprehensive phenotyping: 1) objective physical activity measurement using accelerometers over two weeks; 2) continuous blood glucose monitoring for two weeks, including two standardized test meals, alongside traditional dietary assessment via Food Frequency Questionnaires (FFQ) and 24-hour recalls; 3) assessment of cognitive function and brain imaging using the Addenbrooke's Cognitive Examination-Revised (ACE-R) and brain MRI; and 4) gut microbiome profiling analysis using sequencing techniques.

ELIGIBILITY:
Inclusion Criteria:

Participants from the Guangzhou Nutrition and Health Study, lived in Guangzhou, China, and aged 45 years or older;

Exclusion Criteria:

Metal implants and other contraindications for magnetic resonance imaging scanning

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1425 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2025-04-28 (Actual); Study Completion 2025-05-21 (Actual)

PRIMARY OUTCOMES:
Continuous blood glucose profile over 2 weeks | at enrollment
  Glucose levels were measured by a continuous glucose monitor over 2 weeks.
Brain images | at enrollment
  Brain structure and function were measured by brain magnetic resonance imaging (MRI).

SECONDARY OUTCOMES:
Cognitive scores | at enrollment
  Cognitive function was measured by the Addenbrooke's Cognitive Examination-Revised (ACE-R). The original 26 components were combined to produce five subscores, 100 in total. The cutoff for dementia is 82-88/100.
Incidence of Alzheimer's disease (AD) | 6 and 10 years after enrollment
  New cases of AD will be diagnosed by neurological clinician according to the Chinese guideline for the diagnosis and treatment of Alzheimer's disease dementia(2020).
Structure of gut microbiome profile | At enrollment
  Gut microbiome profile for each participant is measured by metagenome and ITS2 sequencing.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No